CLINICAL TRIAL: NCT06209034
Title: Ultrasonographic Evaluation of Intraoperative Optic Nerve Sheath Diameter Changes in Patients Undergoing Laparoscopic Surgery
Brief Title: Intraoperative Optic Nerve Sheath Diameter Changes After Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sevim Cesur, Associate professor, Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KÜ GOKAEK-2023/19.12
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Optic Nerve Sheath Diameter; Intracranial Pressure Increase
Keywords: Ultrasonography; Optic nerve sheath diameter; Laparoscopic surgery
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Masking Description: Single(Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optic nerve sheath measurement (Other): Optic nerve sheath diameter (ONSD) was detected 3 mm behind the entry point of the optic nerve into the globe in both eyes in each ultrasonographic measurement. ONSD was measured bilaterally 3 mm posterior to the papilla. Transverse measurements were made for each optic nerve.
  Interventions: Other: Optic nerve sheath measurement

INTERVENTIONS:
Other: Optic nerve sheath measurement — ONSD was measured bilaterally 3 mm posterior to the papilla. Transverse measurements were made for each optic nerve.

SUMMARY:
Laparoscopic surgery is a widely used alternative to open surgery; Advantages include reduced bleeding and pain intensity, shorter hospital stay, and improved cosmetic results.

Laparoscopic surgery involves the creation of a carbon dioxide (CO2) pneumoperitoneum to facilitate a clear surgical view, which can result in increased intracranial pressure (ICP).

Ultrasonographic measurement of optic nerve sheath diameter (ONSD) is a simple, non-invasive, yet reliable technique for ICP assessment.Ultrasonographic assessment of optic nerve sheath diameter (ONSD) has been proposed as a non-invasive measurement of intracranial pressure.

DETAILED DESCRIPTION:
Ultrasonographic measurement of optic nerve sheath diameter (ONSD) is a simple, non-invasive, yet reliable technique for ICP assessment. Previous studies have demonstrated that ultrasonographic measurement of ONSD correlates with the degree of ICP and can detect intracranial hypertension in a variety of clinical settings.

It was planned to measure the optic nerve sheath throughout the surgery with the help of a linear ultrasound probe.

Ultrasonographically, in each measurement, the optic nerve sheath diameter (ONSD) was detected 3 mm behind the entry point of the optic nerve into the globe in both eyes. ONSD will be measured bilaterally 3 mm behind the papilla. It will be evaluated by transverse measurement for each optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 aged patients
* American Society of Anesthesiologists Classification (ASA) I-II-III patients
* Patients undergoing laparoscopic surgery

Exclusion Criteria:

* American Society of Anesthesiologists Classification (ASA) IV-V patients
* Those with known ophthalmic disease
* Those with a history of ophthalmic surgery
* Those with any known neurological disorder
* History of intracranial hypertension
* Patients who will undergo open abdominal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of optic nerve sheath diameter | During the operation
  Ultrasound measurement of optic nerve sheath diameter during laparoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Cesur, Study Director — Kocaeli University
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University, Kocaeli
  - Sevim Cesur, Kocaeli